CLINICAL TRIAL: NCT00074048
Title: Phase II Trial Of BL22 Immunotoxin In Hairy Cell Leukemia
Brief Title: BL22 Immunotoxin in Treating Patients Previously Treated With Cladribine for Hairy Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Radhika Parikh, MedImmune Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000341680; NCI-04-C-0014; NCI-6048; NCT00071318 (obsolete NCT alias)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Leukemia
Keywords: refractory hairy cell leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Hairy Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): BL22 immunotoxin
  Interventions: Drug: BL22

INTERVENTIONS:
Drug: BL22 — Dosing via IV on Days 1,3, and 5.

SUMMARY:
RATIONALE: The BL22 immunotoxin can locate tumor cells and kill them without harming normal cells. This may be an effective treatment for hairy cell leukemia that has not responded to treatment with cladribine.

PURPOSE: This phase II trial is studying BL22 immunotoxin to see how well it works in treating patients previously treated with cladribine for hairy cell leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with cladribine-resistant hairy cell leukemia treated with BL22 immunotoxin.

Secondary

* Determine the response duration in patients treated with this drug.
* Determine the safety of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Correlate BL22 blood levels and toxicity of this drug with the development of neutralizing antibodies in these patients.

OUTLINE: Patients receive BL22 immunotoxin IV over 30 minutes on days 1, 3, and 5 followed by rest.

Patients are then evaluated at 8 weeks. Patients achieving complete hematologic remission are followed. All other patients continue to receive BL22 immunotoxin as above on days 1, 3, and 5. Treatment repeats every 4 weeks for up to a total of 16 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR without minimal residual disease (MRD) receive 2 courses beyond CR. Patients achieving CR with MRD receive 4 courses beyond CR.

Patients are followed every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hairy cell leukemia
* CD22-positive disease by fluorescence-activated cell sorting with anti-CD22 antibody
* Meets at least 1 of the following indications for treatment:

  * Absolute neutrophil count less than 1,000/mm^3
  * Hemoglobin less than 10 g/dL
  * Platelet count less than 100,000/mm^3
  * Absolute lymphocyte count greater than 20,000/mm^3
  * Symptomatic splenomegaly
* Meets 1 of the following response criteria:

  * No response
  * Complete response (CR) or partial response (PR) less than 2 years in duration after the last course of prior cladribine
  * CR or PR less than 4 years in duration after a second or later course of prior cladribine

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* AST and ALT no greater than 2.5 times upper limit of normal (ULN)
* Bilirubin no greater than 2.2 mg/dL
* Albumin at least 3.0 g/dL

Renal

* Creatinine no greater than 1.4 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serum that neutralizes more than 75% of the activity of 1 µg/mL of BL22 immunotoxin using a bioassay
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness that would preclude study participation
* Understand and give informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior BL22 immunotoxin
* More than 12 weeks since prior monoclonal antibody therapy

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior systemic cytotoxic chemotherapy

Endocrine therapy

* More than 4 weeks since prior systemic steroids (except stable doses of prednisone no greater than 20 mg/day)

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-10; Primary Completion 2007-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Response rate | After even cycle numbers (2,4,6,8,10)

SECONDARY OUTCOMES:
Duration of Response: [Timeframe: Date that a response begins with the date that PD is documented.] | 30 days after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kreitman, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Matsushita K, Margulies I, Onda M, Nagata S, Stetler-Stevenson M, Kreitman RJ. Soluble CD22 as a tumor marker for hairy cell leukemia. Blood. 2008 Sep 15;112(6):2272-7. doi: 10.1182/blood-2008-01-131987. Epub 2008 Jul 2. PMID 18596230